CLINICAL TRIAL: NCT02466256
Title: Comparison of Intraoperative Performance and Incision Morphology Using Three Injector Devices : Randomized, Clinical Trial
Brief Title: Intra and Postoperative Outcomes With 3 Injectors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Principal Investigator, Abhay R. Vasavada, M.S., F.R.C.S (England), Iladevi Cataract and IOL Research Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-005
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Cataract
Keywords: Intraocular lens implantation
MeSH Terms: conditions — Cataract | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Autosert Group (Placebo Comparator): Procedure / Surgery : Intraocular lens implantation with Autosert injector
  Interventions: Procedure: Intraocular lens implantation; Device: Autosert Injector
- Royale Group (Placebo Comparator): Procedure / Surgery : Intraocular lens implantation with Royale Injector
  Interventions: Procedure: Intraocular lens implantation; Device: Royale Injector
- Monarch III Injector (Placebo Comparator): Procedure / Surgery : Intraocular lens implantation with Monarch III group
  Interventions: Device: Monarch III Injector

INTERVENTIONS:
Procedure: Intraocular lens implantation — Intraocular lens implantation
  Arms: Autosert Group; Royale Group
Device: Autosert Injector — Motorised injection device for intraocular lens implantation
  Arms: Autosert Group
Device: Royale Injector — Manual, plunger type injection device for intraocular lens implantation
  Arms: Royale Group
Device: Monarch III Injector — Manual, screw type injection device for intraocular lens implantation
  Arms: Monarch III Injector

SUMMARY:
This randomized clinical trial compares subjective performance during Intraocular lens (IOL) implantation, as well as incision enlargement and anterior segment morphology on OCT when IOL implantation was performed during microcoaxial phacoemulsification through a 2.2mm incision using one of three injectors :

Manual screw type (Monarch III), Manual plunger type (Royale) and motorised injector (Autosert). Further, the investigators also looked at incision integrity by comparing ingress of trypan blue from the ocular surface into the anterior chamber.

DETAILED DESCRIPTION:
In this randomized, clinical trial, three types of injectors were compared :

1. Manual, screw type injector (Monarch III)
2. Manual, plunger type injector (Royale, ASICO)
3. Motorized injector (Autosert, Alcon)

Having performed a phacoemulsification through 2.2mm incision, IOL implantation was performed using a D cartridge and one of three injectors which was decided in a randomized fashion.

The investigators evaluated incision enlargement at following points : at the end of phacoemulsification, and then, at the end of IOL implantation The investigators also looked at trypan blue ingress into the anterior chamber from the ocular surface. At 1 day, 1 week, and 1 month after surgery anterior segment OCT morphology was also studied.

further, the surgeon was asked to subjectively grade the ease of implantation with each injector

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing phacoemulsification for age-related uncomplicated cataracts through a 2.2mm incision.
* Nuclear or corticonuclear of grade 2 to 4 according to the Lens Opacities Classification System (LOCS III)

Exclusion Criteria:

* Glaucoma,
* uveitis,
* shallow anterior chamber (depth <2.1mm),
* prior ocular trauma or surgery,
* maximal pupillary dilatation <6mm,
* high myopia (axial length >25mm),
* posterior polar cataracts,
* dense cataracts, and
* an IOL power <19.0 D or >25.0 D

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incision enlargement in mm | 1 minute after surgery

SECONDARY OUTCOMES:
Trypan Blue ingress into the anterior chamber in log units | 1 minute after surgery
Incision morphology - qualitative | 1 day, 1 week and 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: abhay r vasavada, ms, frcs, Principal Investigator — iladevi cataract & iol research centre